CLINICAL TRIAL: NCT05625230
Title: Testing the Efficiency of a Psychological Treatment for the Rehabilitation of Action Cognition in Depression
Brief Title: Treatment for Rehabilitation of Action Cognition in Depression
Acronym: T-RAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oradea (Other)
Collaborators: York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN-III-P1-1.1-TE-2021-1090
Record Dates: First submitted 2022-11-09; First posted 2022-11-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-11

CONDITIONS: Depression
Keywords: Depression; Behavioural Activation; Dynamic Imagery; Kinect
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors are blind to the conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior activation-PLUS T-RAC (Experimental): Behavioral: Behavior activation/BA plus T-RAC Each session is focused on reviewing the activity log, planning anti-depressant activities for the next week, and finding support for the implementation of the activity. After activity planning, the participants will follow an XboxKinect exergame for 10 minutes, an actfulness exercise and will imagine one planned activity using dynamic imagery. From session 2 restructuring action memories are added.
  Interventions: Behavioral: Behavioral Activation plus Dynamic Mental Imagery
- Arm 2 Behavioral activation (Active Comparator): Behavioral: Behavior activation/BA Participants in the behavioral activation arm will undergo a BA procedure. A therapist will administer an 8 sessions behavioral activation intervention based on the manual used in the COBRA trial.
  Each session is focused on reviewing the activity log, planning anti-depressant activities for the next week, and finding support for the implementation of the activity.
  Interventions: Behavioral: Behavioral activation

INTERVENTIONS:
Behavioral: Behavioral Activation plus Dynamic Mental Imagery — This intervention consists of an 8-session behavioural activation treatment with an added dynamic imagery exercise after each session. The dynamic imagery exercise is structured as follows: (1) the therapist explains the intervention; (2) the therapist models dynamic simulation skill (dynamic imagery) and repeats with the participant while giving appropriate feedback; (3) the participant completes a 10-minute Kinect training; (4) the participant completes a short Actfulness exercise that involves focusing on the feelings of movements of breathing and hands and dynamic imagery of one planned activity. From the second session, participants memorize daily activities forming a short dynamic memory of the activity focusing on feelings of movements.
  Arms: Behavior activation-PLUS T-RAC
Behavioral: Behavioral activation — The BA intervention is a short 8 session behavioural intervention. Participants learn to monitor the activities, plan "anti-depressant" activities for the next week and find support for the implementation of the activity.
  Arms: Arm 2 Behavioral activation

SUMMARY:
The present research study investigates the effects of a brief dynamic imagery intervention added to a short behavioral activation treatment on the treatment acceptability, feasibility, and primary efficacy for individuals with depression. Behavioral activation treatment is a standard treatment for depression. To enhance behavioral activation treatment acceptance and efficacy, a dynamic imagery intervention was added to augment the motor component of imagery and memories. Two types of treatment were compared: (1) behavioral activation treatment and (2) behavioral activation treatment plus dynamic imagery. The behavioral activation treatment is a short 8-session intervention based on a dynamic imagery procedure for enhancing the recruitment of motor activation in cognitive processing. 110 participants will be randomized into two groups. Half will be randomized to standard behavioral activation treatment and a half to behavioral activation treatment plus imagery treatment. Participants complete the assessment before, during (weekly), and after treatment. Follow-up will be measured at 3 months after the end of the treatment.

DETAILED DESCRIPTION:
Major depressive disorder is a highly prevalent and chronic disorder incurring significant costs to society. Although several treatments are recommended for the treatment of major depressive disorder, the high rate of recurrence suggests the need for constant improvement in the treatments for depression. Cognitive deficits following depressive episodes are possible targets to improve existing treatments. Cognitive symptoms are residual symptoms and often interfere with the ability of individuals with depression to solve life problems. Building on the idea that action cognition and motor imagery deficits are more stable in depressed individuals a rehabilitation-type of motor imagery training was developed. It is based on principles of rehabilitation of motor imagery (used in sport as in the field of neurorehabilitation), for individuals with neurological conditions. It does integrate a forward modeling of action and motor imagery, remote kinematics (Kinect) and embodied cognition account. This new intervention proved efficient in clinical work. There are several steps to the intervention. In the first session, the therapist explains the intervention and teaches a dynamic simulation routine. Then, the patient undergoes Kinect training for 10 minutes followed by an actfulness exercise focusing on feelings of movement that focuses on sensations of movement and dynamic imagining of a planned activity. In the second session, patients are thought to restructure action memories. The intervention is based on the scaffolding of two well-known interventions: mindfulness meditation-movement meditations and memory restructuring. Deficient action simulations are rehabilitated by: (a) partial movements (alternating covert with dynamic-partial movements simulations in response to stimuli); (b) linguistic supports (training in gerundival perceptions, e.g., recognize and naming a stimuli by actions, e.g., a door to open), (c) enhanced perceptual and affective simulations and (d) episodic memory support (participants have to form future memories of action cores-last sequence of movement before the perception of desired environmental change, correct them by experience and remember at the end of the day). Thus, it is a rehearsal training including combined actual and mental practice with augmentation of the motor component of simulations in thinking by enhancing gestures, language and episodic memory as controls of simulation, and is applied to promote the use of motor simulations in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken Romanian
* Reporting clinically significant depressive symptoms above cut-off on depression measures and by structured clinical interview

Exclusion Criteria:

* Elevated risk of suicide/Suicide intent and plans
* Current substance use disorder
* Current or previous manic/hypomanic episodes
* Current psychotic disorder
* Current diagnosis of dementia/major neurocognitive disorder
* Currently receiving psychological therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms severity measured by Beck Depression Inventory II, | Baseline; Intervention Week 8; 3 months post-intervention
  Beck Depression Inventory II is a 21-item questionnaire used to measure severity of depression. The score ranges from 0-63. Higher scores indicate higher depression.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms using the Patient Health Questionnaire 9 | Baseline; Intervention Week 1; Intervention Week 2; Intervention Week 3; Intervention Week 4; Intervention Week 5; Intervention Week 6; Intervention Week 7; Intervention Week 8; 3 months post-intervention
  Patient Health Questionnaire 9 is a nine-item questionnaire used to identify depression as well as measuring severity of depression. The score ranges from 0-27. Higher scores indicate higher severity of depression.
Change from baseline in anhedonia symptoms using the Snaith-Hamilton Pleasure Scale | Baseline; Intervention Week 8; 3 months post-intervention
  Snaith-Hamilton Pleasure Scale is a 14-item questionnaire used to measure anhedonia. The score ranges from 0-14. Higher scores indicate higher anhedonia.
Changes from baseline in apathy level using Motivational Apathy Index | Baseline; Intervention Week 8; 3 months post-intervention
  Motivational Apathy Index is an 18-item questionnaire used to identify three dimensions of apathy assessed with the mean score, which ranges from 0-4. Higher scores indicate higher apathy.
Change from baseline in the diagnosis of depression assessed using the Structured Clinical Interview for DSM-5 Disorders -- Clinician Version | Baseline; Intervention Week 8
  Structured Clinical Interview for DSM-5 Disorders is a structured clinical interview used to assess the presence/absence of common psychiatric disorders.
Change from baseline in the health and disability level using The WHO Disability Assessment Schedule 12-item | Baseline; Intervention Week 8; 3 months post-intervention
  he WHO Disability Assessment Schedule 12-item is a 12-item questionnaire used to assess disability due to health conditions. The total score ranges from 0-48. Higher scores indicate higher functioning.
Scores for adverse and unwanted effects of the experimental intervention | Week 8
  Negative incidents and effects of psychological treatment scale is a 20-item questionnaire used to assess adverse and unwanted effects of psychological treatments. The total score ranges from 0-80. Higher scores indicate higher negative effects.
Change from baseline in the motor imagery is assessed at baseline using the Vividness of Motor Imagery Questionnaire-2 | Baseline; Intervention Week 6
  Vividness of Motor Imagery Questionnaire-2 is a 12-item questionnaire assessing the vividness of mental imagery. It has three subscales, each subscale having a total score ranging from 12-60. Higher scores indicate lower vividness of imagery.
Change from baseline in affect and behaviour monitoring scale | Baseline; Intervention Week 1; Intervention Week 2; Intervention Week 3; Intervention Week 4; Intervention Week 5; Intervention Week 6; Intervention Week 7; Intervention Week 8; 3 months post-intervention
  The affect and behavior monitoring scale is 7-point Likert scale built for the present study to monitor weekly changes in functioning emotions, behaviour profile, efficacy, difficulty of simulation. For each item, the score ranges from 1 to 7. Higher scores mean higher functioning.
Change from baseline in the Environmental and Reward Observation Scale | Baseline; Intervention Week 6
  The Environmental and Reward Observation Scale is a 10-item scale assessing the level of rewards. The total score ranges from 10-40. Higher scores indicate higher rewards.
Change from baseline in the rumination style scale | Baseline; Intervention Week 6
  The Rumination Style Scale scale is a short 10 item scale that measure the level of rumination. Scores ranges from a low of 14 to a high of 40. Higher scores indicate higher difficulties with rumination.
Change from baseline in the behavioral activation level using The Behavioral Activation for Depression Scale - Short Form | Baseline; Intervention Week 6; Intervention Week 8
  The Behavioral Activation for Depression Scale is a nine-item questionnaire used to measure changes in avoidance and activation. The score ranges from 0-54. Higher scores indicate higher avoidance.
Change from baseline in Backward digit span task | Baseline; Intervention Week 6 Intervention Week 8
  In the Backward digit span task, participants are given a series of digits and asked to repeat them backward. The score is how many numbers of participants repeat backward. A higher score indicates better working memory
Change from baseline in verbal fluency task | Baseline; Intervention Week 6; Intervention Week 8
  In the verbal fluency task participants must generate as many words as possible starting with a consonant (F, S or T) in one minute. The score is the number of words in one minute for one letter. A higher score indicates better verbal fluency.
Change from baseline in verb fluency task | Baseline; Intervention Week 6; Intervention Week 8
  The verb fluency task asks participants to generate as many verbs as possible in one minute. The score is the number of verbs generated in one minute. A higher score indicates better verb fluency.
Change from baseline in anxiety symptoms using the Generalized Anxiety Disorder 7-item | Baseline; Intervention Week 8
  Generalized Anxiety Disorder 7 is a seven-item questionnaire used to identify generalized anxiety disorder as well as measuring severity of anxiety symptoms. The score ranges from 0-21. Higher scores indicate higher severity of anxiety.
Change from baseline in The Movement Imagery Questionnaire-3 | Baseline; Intervention Week 6
  The Movement Imagery Questionnaire-3 is a questionnaire consisting of total of 12 items to assess individual's ability to image four movements. It has two visual scales and a kinesthesic scale, scores range for each scale from 4 to 28 with a higher score representing a better mental imagery ability.
Acceptability ratings | Week 8
  For acceptability ratings, the participants rate on a 5-points Likert scale their satisfaction, intention to continue and to recommend the intervention. Higher score means higher acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Tiba, PhD, Study Director — University of Oradea
Locations (1):
- University of Oradea, Oradea, Bihor County, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From June/July 2023

REFERENCES:
- [Background] Martell, Christopher R., Sona Dimidjian, and Ruth Herman-Dunn. Behavioral activation for depression: A clinician's guide. Guilford Publications, 2021.
- [Background] Ang YS, Lockwood P, Apps MA, Muhammed K, Husain M. Distinct Subtypes of Apathy Revealed by the Apathy Motivation Index. PLoS One. 2017 Jan 11;12(1):e0169938. doi: 10.1371/journal.pone.0169938. eCollection 2017. PMID 28076387
- [Background] Beshai S, Dobson KS, Bockting CL, Quigley L. Relapse and recurrence prevention in depression: current research and future prospects. Clin Psychol Rev. 2011 Dec;31(8):1349-60. doi: 10.1016/j.cpr.2011.09.003. Epub 2011 Sep 17. PMID 22020371
- [Background] Bortolato B, Miskowiak KW, Kohler CA, Maes M, Fernandes BS, Berk M, Carvalho AF. Cognitive remission: a novel objective for the treatment of major depression? BMC Med. 2016 Jan 22;14:9. doi: 10.1186/s12916-016-0560-3. PMID 26801406
- [Background] Chen J, Yang LQ, Zhang ZJ, Ma WT, Wu XQ, Zhang XR, Wei DH, Fu QH, Liu GX, Deng ZH, Hua Z, Zhang Y, Jia T. The association between the disruption of motor imagery and the number of depressive episodes of major depression. J Affect Disord. 2013 Sep 5;150(2):337-43. doi: 10.1016/j.jad.2013.04.015. Epub 2013 May 16. PMID 23684121
- [Background] Gorwood P, Richard-Devantoy S, Bayle F, Clery-Melin ML. Psychomotor retardation is a scar of past depressive episodes, revealed by simple cognitive tests. Eur Neuropsychopharmacol. 2014 Oct;24(10):1630-40. doi: 10.1016/j.euroneuro.2014.07.013. Epub 2014 Aug 2. PMID 25129432
- [Background] Shadmehr R, Smith MA, Krakauer JW. Error correction, sensory prediction, and adaptation in motor control. Annu Rev Neurosci. 2010;33:89-108. doi: 10.1146/annurev-neuro-060909-153135. PMID 20367317
- [Background] Glenberg AM. Embodiment as a unifying perspective for psychology. Wiley Interdiscip Rev Cogn Sci. 2010 Jul;1(4):586-596. doi: 10.1002/wcs.55. Epub 2010 Apr 8. PMID 26271505
- [Background] Tiba A, Voss L. A motor imagery training for improving action cognition results in the reduction of residual symptoms after major depressive disorder: a single case study. Journal of Evidence- Based Psychotherapies. 2022: Vol. 22, No. 1, March 2022, 137- 168./ 10.24193/je bp.2022.1.8
- [Background] Holmes PS, Collins DJ. The PETTLEP Approach to Motor Imagery: A Functional Equivalence Model for Sport Psychologists. Journal of Applied Sport Psychology. 2001: 13:1, 60-83, DOI: 10.1080/10413200109339004
- [Background] Courtine G, Papaxanthis C, Gentili R, Pozzo T. Gait-dependent motor memory facilitation in covert movement execution. Brain Res Cogn Brain Res. 2004 Dec;22(1):67-75. doi: 10.1016/j.cogbrainres.2004.07.008. PMID 15561502
- [Background] Malouin F, Jackson PL, Richards CL. Towards the integration of mental practice in rehabilitation programs. A critical review. Front Hum Neurosci. 2013 Sep 19;7:576. doi: 10.3389/fnhum.2013.00576. PMID 24065903
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] First B, Williams JB, Karg RS, Spitzer RL. Structured Clinical Interview for DSM-5 Disorders, Clinician Version (SCID-5-CV) 2015: Arlington, VA: American Psychiatric Association.
- [Background] Manos RC, Kanter JW, Luo W. The behavioral activation for depression scale-short form: development and validation. Behav Ther. 2011 Dec;42(4):726-39. doi: 10.1016/j.beth.2011.04.004. Epub 2011 Jun 1. PMID 22036000
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Callow N, Roberts R. Imagery research: An investigation of three issues. Psychology of Sport & Exercise.2010: 11, 325-329.
- [Background] Armento ME, Hopko DR. The Environmental Reward Observation Scale (EROS): development, validity, and reliability. Behav Ther. 2007 Jun;38(2):107-19. doi: 10.1016/j.beth.2006.05.003. Epub 2006 Dec 12. PMID 17499078
- [Background] Treynor W, Gonzalez R, Nolen-Hoeksema S. Rumination reconsidered: a psychometric analysis. Cogn Ther Res. 2003;27(3):247-59.
- [Background] Martell CR, Addis ME, Jacobson NS. Depression in context: Strategies for guided action. 2001: W W Norton & Co.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440